CLINICAL TRIAL: NCT02229890
Title: SITS-NEW Safe Implementation of Thrombolysis in Stroke in the Non EU-World: An International Observational Study of the Safety and Efficacy of Thrombolysis in Stroke
Brief Title: An International Observational Study of the Safety and Efficacy of Thrombolysis in Stroke
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 135.317
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Acute ischemic stroke within three hours after symptom onset
  Interventions: Drug: alteplase

INTERVENTIONS:
Drug: alteplase
  Other Names: Actilyse®

SUMMARY:
Study to evaluate the safety and efficacy of intravenous recombinant tissue Plasminogen Activator, alteplase, Actilyse® (rt-PA) (0.9 mg/kg) within 3 hours of symptom onset in acute ischemic stroke

ELIGIBILITY:
Inclusion Criteria:

* Female or male inpatients
* Age 18 - 80 years
* Clinical diagnosis of ischemic stroke causing a measurable neurological deficit defined as impairment of language, motor function, cognition, gaze, vision and/or neglect. Ischemic stroke is defined as an event characterized by sudden onset of acute focal neurological deficit, presumed to be caused by cerebral ischemia, after CT scan exclusion of hemorrhage
* Onset of symptoms within 3 hours prior to initiation of thrombolysis treatment
* Stroke symptoms present for at least 30 minutes and not significantly improved before treatment. Symptoms must be distinguishable from an episode of generalized ischemia (i.e. syncope), seizure, or migraine disorder
* Patients are willing to receive thrombolysis treatment and to give informed consent with regard to retrieval and storage of data and follow up procedures, according to the regulations in participating countries
* Willingness and ability to comply with the observational study protocol

Exclusion Criteria:

* Evidence of intracranial hemorrhage (ICH) on the CT-scan.
* Symptoms of ischemic attack began more than 3 hours prior to infusion start or when time of symptom onset is unknown
* Symptoms of acute ischemic stroke that were either rapidly improving or only minor before start of infusion
* Severe stroke as assessed clinically and/or by appropriate imaging techniques
* Seizure at onset of stroke
* History of previous stroke or serious head-trauma within three months
* Administration of heparin within the previous 48 hours preceding the onset of stroke with an elevated activated thromboplastin time (aPTT) at presentation
* A combination of previous stroke and concomitant diabetes
* Platelet count of below 100,000/mm³
* Systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg, or aggressive management (repeated IV medication) necessary to reduce BP to these limits.
* Blood glucose <50 or > 400 mg/dl
* Significant bleeding disorder at present or within the past 6 months, known hemorrhagic diathesis
* Patients receiving oral anticoagulants, e.g. warfarin sodium (INR>1.3)
* History or evidence or suspicion of intracranial hemorrhage including sub-arachnoid hemorrhage
* Severe uncontrolled arterial hypertension
* Any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery)
* Hemorrhagic retinopathy, e.g. in diabetes (vision disturbances may indicate hemorrhagic retinopathy) or other hemorrhagic ophthalmic conditions
* Bacterial endocarditis, pericarditis
* Prolonged or traumatic cardiopulmonary resuscitation (>2 minutes), obstetrical delivery within the past 10 days, recent puncture of a non-compressible blood-vessel (e.g. subclavian or jugular vein puncture)
* Acute pancreatitis
* Documented ulcerative gastrointestinal disease during the last 3 months
* Arterial aneurysm, arterial/venous malformation
* Neoplasm with increased bleeding risk
* Severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension (oesophageal varices) and active hepatitis
* Major surgery or significant trauma in past 10 days (this includes any trauma associated with current acute myocardial infarction), recent trauma to head or cranium
* Hypersensitivity to the active substance alteplase or to any of the excipients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke within three hours after symptom onset treated at stroke centers
Sampling Method: Non-Probability Sample
Enrollment: 593 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of symptomatic intracerebral hemorrhage (Cochrane definition) | up to 7 days
Occurrence of symptomatic intracerebral hemorrhage (SITS-MOST definition) | up to 36 hours
Mortality rate | up to 6 months

SECONDARY OUTCOMES:
Number of patients with functional independence (independence for activities of daily living) | 3 months
  Rankin score 0-2